CLINICAL TRIAL: NCT04771949
Title: Prevalence and Environmental Risk Indicators for Periodontitis. A Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Researcher, University of Siena
Other Study IDs: LF001
Record Dates: First submitted 2021-02-16; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Periodontal Diseases; Periodontitis; Lifestyle; Mediterranean Diet
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients coming to the University Clinic of Dentistry: All patients coming to the dental University Clinic will be screened for the inclusion in the study.
  Interventions: Diagnostic Test: Full periodontal chart; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: Full periodontal chart — A full periodontal chart will be carried out including all biometric periodontal variables: Probing Pocket Depth (PPD), Bleeding on Probing (BoP), presence of Plaque, recession (REC), Full Mouth Plaque Score (FMPS), Full Mouth Bleeding Score (FMBS), presence of furcation and mobility. Periodontal status, as assessed by the periodontal chart, will be evaluated following the New Classification of Periodontal and Peri implant diseases.
Other: Questionnaires — After the periodontal chart, patients will be administered the italian version of 4 questionnaires regarding:
  1. Adherence to Mediterranean Diet (Gnagnarella et al. 2018);
  2. International Physical Activity Questionnaire (IPAQ) (Mannocci et al. 2010);
  3. Pittsburgh Sleep Quality Index (PSQI) (Curcio et al. 2013);
  4. Italian Perceived Stress Scale (Fossati, 2010).

SUMMARY:
Periodontitis is a biofilm-mediated chronic inflammatory disease with a multi-factorial etiology; it belongs to the group of diseases classified as "Non-communicable Diseases" (NCDs). According to the results of the Global Burden of Disease Study of 2017, it is the sixth most prevalent disease worldwide and it constitutes a heavy burden on health costs.

Risk factors for such disease include non-modifiable risk factors, i.e. familiarity, diabetes, cardiovascular diseases, metabolic syndrome, as well as modifiable risk factors, i.e. diet, stress and low physical exercise. Given the significant impact of oral health on the quality of life and overall well being of the individual, many studies investigated the importance of risk factors for oral health. In particular, there is some evidence that more severe manifestations of periodontitis are associated with lower physical activity (De Oliveira Ferreira et al., 2019), poor sleep quality (Karaaslan & Dikilitaş, 2019) and more perceived stress (Coelho et al., 2020). With regards to diet, despite the high number of studies demonstrating an anti-inflammatory effect of the Mediterranean Diet, no study has ever investigated the adherence to Mediterranean Dieta to the oral health status.

From a methodological standpoint, investigations regarding environmental factors are mainly carried out through questionnaires administration, whose validity and reproducibility had been previously demonstrated. The novelty introduced by the present study would be a complete analysis of the effects of lifestyles (diet, sleep quality, physical exercise, perceived stress) on the periodontal status of the individual.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years old;
* ability and willingness to give informed consent.

Exclusion Criteria:

* pregnancy or lactation;
* inability to communicate either in English or Italian;
* inability or unwillingness to give informed consent.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients coming to the dental University clinic will be screened for the inclusion in the study
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-11-18 (Estimated); Study Completion 2021-11-29 (Estimated)

PRIMARY OUTCOMES:
Prevalence of periodontitis | Baseline
  The prevalence of periodontitis among a sample of patients coming to the dental University clinic will be calculated

SECONDARY OUTCOMES:
Adherence to mediterranean diet | Baseline
  The secondary aim will be to relate the presence and severity of periodontitis to the adherence to Mediterranean diet, measured through a questionnaire (Gnagnarella et al. 2018) on a scale between 0 to 9. The higher the score, the higher the adherence to Mediterranean diet.
Sleep Quality | Baseline
  The secondary aim will be to relate the presence and severity of periodontitis to sleep quality, measured through a questionnaire (Pittsburgh Sleep Quality Index) on a scale between 0 to 21. The higher the score, the poorer the sleep quality.
Physical Activity | Baseline
  The secondary aim will be to relate the presence and severity of periodontitis to the amount of physical exercise, measured through a questionnaire (International Physical activity questionnaire, IPAQ) on a scale between 0 to 2 (0= low physical activity; 1= moderate physical activity; 2= intense physical activity)
Italian Perceived Stress Scale (IPSS) | Baseline
  The secondary aim will be to relate the presence and severity of periodontitis to the amount of stress perceived, measured through a questionnaire (Italian perceived stress scale) on a scale between 0 to 40. The higher the score, the higher the amount of stress perceived.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy